CLINICAL TRIAL: NCT03122743
Title: Correlation of Serum Catecholamine With Emotional Stress in Men With Prostate Cancer: A Pilot Study
Brief Title: Collection of Serum Samples in Studying Emotional Stress in Patients With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00041151; NCI-2016-01590 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 85316 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-10-27; First posted 2017-04-21 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Hormone-Resistant Prostate Cancer; Recurrent Prostate Carcinoma; Stage I Prostate Cancer; Stage II Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (collection of samples, questionnaires): Patients undergo collection of serum samples for epinephrine and cortisol levels at baseline and 4 clinical visits. Patients also receive the Self-Perceived Stress questionnaire and the Distress Thermometer questionnaire to measure perceived stress.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of serum samples
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot research trial studies the collection of serum samples in studying emotional stress in patients with prostate cancer. Studying serum samples from patients with prostate cancer in the laboratory may help doctors determine if levels of epinephrine and cortisol, substances the body makes when stressed, rise or fall with how patients are feeling and/or if those levels are related to clinical information related to prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if serum epinephrine or cortisol levels in men with prostate cancer correlate with perceived stress or distress over time in two to five consecutive visits.

SECONDARY OBJECTIVES:

I. To determine the change in serum epinephrine levels in men with prostate cancer over time in two to five consecutive visits.

II. To determine the change in serum cortisol levels in men with prostate cancer over time in two to five consecutive visits.

III. To determine the change in levels of stress in men with prostate cancer over time in two to five consecutive visits IV. To determine the change in levels of distress in men with prostate cancer over time in two to five consecutive visits.

TERTIARY OBJECTIVES:

I. To determine if serum epinephrine or cortisol levels in men with prostate cancer correlate with prostate cancer progression two to five visits.

OUTLINE:

Patients undergo collection of serum samples for epinephrine and cortisol levels at baseline and 4 clinical visits. Patients also receive the Self-Perceived Stress questionnaire and the Distress Thermometer questionnaire to measure perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2
* Individuals able to understand and willing to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* History of current or past medical or psychiatric illness that would make participation difficult or not feasible at the discretion of the principal investigator or co-investigators

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Change in distress score, assessed by the Distress Thermometer | Up to 1 year
  Will calculate the patient's stress levels at each of the 5 visits using a validated distress thermometer
Change in perceived stress scores, assessed by the Self-Perceived Stress Questionnaire | Up to 1 year
  Will calculate the patient's stress levels at each of the 5 visits using a validated measure of self-perceived stress
Change in serum cortisol levels | Up to 1 year
  Will calculate the change in serum cortisol levels between the first and last assessment and calculate the corresponding change in perceived stress or distress during the same time period. Will estimate the Pearson correlation between the two changes. Will also estimate a 95% confidence interval for this estimated correlation. These calculations will be performed overall (pooling all 3 groups together) and then repeated for each of the three groups of men separately. Will fit a longitudinal mixed model that incorporates the repeated measures taken on each patient. Additional int
Change in serum epinephrine levels | Up to 1 year
  Will calculate the change in serum epinephrine levels between the first and last assessment and calculate the corresponding change in perceived stress or distress during the same time period. Will estimate the Pearson correlation between the two changes. Will also estimate a 95% confidence interval for this estimated correlation. These calculations will be performed overall (pooling all 3 groups together) and then repeated for each of the three groups of men separately. Will fit a longitudinal mixed model that incorporates the repeated measures taken on each patient. Additional int

SECONDARY OUTCOMES:
Change in levels of distress assessed by the Distress Thermometer | Baseline up to 1 year
  Will fit a two-way random effects model to examine the time course of distress levels.
Change in self-perceived stress, assessed by the Self-Perceived Stress Questionnaire | Baseline up to 1 year
  Will fit a two-way random effects model to examine the time course of stress levels.
Change in serum cortisol levels | Baseline up to 1 year
  Will fit a two-way random effects model to examine the time course of serum cortisol levels.
Change in serum epinephrine levels | Baseline up to 1 year
  Will fit a two-way random effects model to examine the time course of serum epinephrine levels.

OTHER OUTCOMES:
Change in levels of serum prostate specific antigen in patients with complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) | Baseline up to 1 year
  Will determine whether there are any differences at each of the time points in serum epinephrine or cortisol levels using one-way analysis of variance (ANOVA) models.
Change in serum cortisol AUC values | Baseline up to 1 year
  Will be compared across the 4-levels of progression (CR, PR, SD, and PD) or 2-levels of progression (CR/PR vs SD/PD) using ANOVA models. These models can be run separately for each of the 3 groups of patients - and also in an overall model with all patients included and a covariate for group and group by AUC value interaction.
Change in serum epinephrine area under the curve (AUC) values | Baseline up to 1 year
  Will be compared across the 4-levels of progression (CR, PR, SD, and PD) or 2-levels of progression (CR/PR vs SD/PD) using ANOVA models. These models can be run separately for each of the 3 groups of patients - and also in an overall model with all patients included and a covariate for group and group by AUC value interaction.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Frizzell, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT03122743/ICF_000.pdf